CLINICAL TRIAL: NCT05434442
Title: Evaluation of the Effectiveness of the Simulation Model and Mobile Application in Teaching Tracheostomy Aspiration Application to the Caregivers of Patients With Tracheostomy and Tracheotomy
Brief Title: Caregivers Tracheal Aspiration Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Yeliz Sapulu Alakan, Lecturer, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Uludag Universty
Record Dates: First submitted 2022-06-14; First posted 2022-06-28 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Tracheostomy; Family Caregivers; Aspiration
Keywords: Family Caregivers; Tracheostomy aspiration; Mobile application; Simulation training
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Caregivers will be assigned to control, simulation and mobile application groups by block randomization method. An equal number of caregivers from each clinic will be assigned to each group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Caregivers will be assigned to control, simulation and mobile application groups by block randomization method, and communication between groups will be controlled. Caregivers assigned to groups by block randomization method will be numbered. Skill evaluation videos will be taken by a researcher. Skill assessments will also be made by another blinded researcher to the groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1-simulation model training (Other): Tracheal aspiration training of caregivers assigned to the "simulation training group" will be given to the same standard by researcher. It will be shown in practice on the tracheostomy care simulator. They will also receive clinical routine training
  Interventions: Other: simulation model training; Other: control group
- 2-mobile app training (Other): An animation-based mobile application will be installed on the phones of the caregivers assigned to the "mobile application group" and will be introduced and made available to their use by the researcher. They will also receive clinical routine training
  Interventions: Other: mobile app training; Other: control group
- 3-control group (Other): Clinical routine training will be given to caregivers in this group.
  Interventions: Other: control group

INTERVENTIONS:
Other: simulation model training — Tracheal aspiration training of caregivers assigned to the "simulation training group" will be given to the same standard by researcher. It will be shown in practice on the tracheostomy care simulator.
  Arms: 1-simulation model training
Other: mobile app training — An animation-based mobile application will be installed on the phones of the caregivers assigned to the "mobile application group" and will be introduced and made available to their use by the researcher.
  Arms: 2-mobile app training
Other: control group — Clinical routine training will be given to caregivers in this group.

SUMMARY:
The aim of this study is to determine the effects of animation-based mobile application and simulation-based training methods on tracheal aspiration knowledge and skills of patient relatives who care for patients with tracheostomy/tracheotomy. Experimental pre-test-post-test control group study design was planned.

DETAILED DESCRIPTION:
The study aims to determine the effect of tracheal aspiration training given to caregivers of patients with tracheostomy and tracheotomy. The effects of training given using clinical routine training, animation-based mobile application and simulation-based training methods on the knowledge and skills of caregivers will be evaluated. Experimental pre-test-post-test control group study design was planned. This study will be carried out as a multicenter in Bursa, Turkey.The centers where the study will be conducted are Bursa Uludağ University Health Research and Application Center and Bursa City Hospital. In calculating the sample size, the effect size was determined as 0.4 for 80% power and 5% significance level. In this direction, it is aimed to include 22 patient relatives in each group in order to compare the knowledge and skill levels between the mobile application, simulation training and control groups. A total of 66 patient relatives will be included in the study. The caregivers to be assigned to the groups will be selected using the block randomized method.

The plan to be implemented in the research;

1. Pre-Training: "Introductory Characteristics Form" and "Information Evaluation Form" will be filled in for caregivers in all groups.
2. Training: An animation-based mobile application will be installed on the phones of the caregivers assigned to the "mobile application group" and will be introduced and made available to their use by the researcher Yeliz ŞAPULU ALAKAN.

   Tracheal aspiration training of caregivers assigned to the "simulation training group" will be given to the same standard by researcher Yeliz ŞAPULU ALAKAN. It will be shown in practice on the tracheostomy care simulator.

   Caregivers assigned to the "control group" will not undergo any training other than routine in-clinic training on tracheostomy aspiration.

   Caregivers in the all group will also undergo routine training of the clinic
3. After the training: Caregivers in all groups will fill out the "Training Evaluation Form" and "Information Evaluation Form." The video of the caregiver taken during the tracheal aspiration procedure will be evaluated by the researchers using the "Skill Evaluation Form".
4. One month after the training: Caregivers in all groups will fill in the "Information Evaluation Form" and "Result Evaluation Form".The video of the caregiver taken during the tracheal aspiration procedure will be evaluated by the researchers using the "Skill Evaluation Form".

ELIGIBILITY:
Inclusion Criteria:

* Being the primary caregiver of the patient who will undergo a tracheotomy or tracheostomy, which is expected to last at least one month,
* Primary care will be continued by the same caregiver for a period of one month.
* Volunteering to participate in the research
* Being over 18 years old,
* Absence of a diagnosed psychiatric illness that may interfere with communication
* Owning and being able to use a smart mobile phone

Exclusion Criteria:

* Not being the primary caregiver of the patient who will undergo tracheostomy or tracheotomy,
* Change of primary caregiver in less than a month
* Closing the tracheotomy in less than a month
* Not volunteering to participate in the research
* Be under the age of 18,
* Having a diagnosed psychiatric illness that may interfere with communication
* Not having or being unable to use a smart mobile phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
To determine the effects of simulation model, mobile application and routine training methods on the knowledge scores of the caregivers of patients with tracheostomy before the training, after the training and one month after the training. | through study completion, an average of 1 year
  Getting at least 50 points from each part of the "knowledge evaluation form", which includes questions about the procedure.
To determine the effects of simulation model, mobile application and routine training methods on the skill levels of caregivers of patients with tracheostomy before, after and one month after training. | through study completion, an average of 1 year
  Caregivers will be evaluated according to the "skill evaluation form" during the aspiration process from the tracheostomy.

SECONDARY OUTCOMES:
Satisfaction with different training methods | through study completion, an average of 1 year
  To be measured using the "Satisfaction Evaluation Form"
One month after the different trainings, the effects of caregivers on the aspiration application will be evaluated using the "Results Evaluation Form". | through study completion, an average of 1 year
  The effect of different training methods will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: yeliz Şapulu Alakan, Principal Investigator — Uludag Universty; Neriman Akansel, Study Director — Uludag Universty
Locations (2):
- Turkey (Türkiye) (2):
  - Yeliz, Bursa, Nilüfer
  - Bursa Uludag university, Bursa

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, CSR
Time Frame: After the research is published
Access Criteria: It will be shared by researcher Yeliz ŞAPULU ALAKAN to be used in meta analysis or other research.

REFERENCES:
- [Background] Bayram SB, Caliskan N. Effect of a game-based virtual reality phone application on tracheostomy care education for nursing students: A randomized controlled trial. Nurse Educ Today. 2019 Aug;79:25-31. doi: 10.1016/j.nedt.2019.05.010. Epub 2019 May 9. PMID 31102793
- [Background] Loerzel VW, Crosby WW, Reising E, Sole ML. Developing the Tracheostomy Care Anxiety Relief Through Education and Support (T-CARES) Program. Clin J Oncol Nurs. 2014 Oct;18(5):522-7. doi: 10.1188/14.CJON.522-527. PMID 25253106
- See also: Guidelines for the Care of Patients with Tracheostomy Tubes — https://www.google.com/search?q=Guidelines+for+the+Care+of+Patients+with+Tracheostomy+Tubes&rlz=1C1CHZN_trTR930TR930&oq=Guidelines+for+the+Care+of+Patients+with+Tracheostomy+Tubes&aqs=chrome..69i57j0i19i22i30.1056j0j7&sourceid=chrome&ie=UTF-8
- See also: A Caregiver Guide for Tracheostomy Care at Home — https://silo.tips/queue/a-caregiver-guide-for-tracheostomy-care-at-home
- See also: Tracheostomy Teachıng Package For Parents And Carers Assessment. — https://mft.nhs.uk/app/uploads/2020/08/Tracheostomy-Teaching-Package-for-Parents-and-Carers.pdf.